CLINICAL TRIAL: NCT06855550
Title: Evaluation of Plasmatic Magnesium Levels and Its Association with Atrial Fibrillation After Cardiac Surgery
Brief Title: Postoperative Incidence of Atrial Fibrillation Following Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Fundación Cardioinfantil Instituto de Cardiología (Other)
Responsible Party: Principal Investigator, Edgar Hernández Leiva, Head of Cardiovascular Critical Care, Fundación Cardioinfantil Instituto de Cardiología
Other Study IDs: 2023PROCCA0043; 2023PROCCA0043 (Other: Fundación Cardioinfantil-Instituto de Cardiología)
Record Dates: First submitted 2025-02-24; First posted 2025-03-04 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation (AF); Hypomagnesemia; Cardiac Surgery
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Postoperative cardiac surgery: Patients who will undergo elective cardiac surgery of any kind will be included, except those with a history of preoperative atrial fibrillation, urgent/emergency surgery, or those who will undergo maze surgery (alone or in combination with other procedures).
  Magnesium levels will be measured immediately after surgery and every subsequent 12-24 hours during the stay in the intensive care unit. Each patient will be followed up, and morbidity and mortality will be recorded through in-hospital evaluation or up to 30 days postoperatively (whichever occurs first). Follow-up will be performed by a member of the research team who will be blinded to the postoperative magnesium levels. Preoperative evaluation, premedication, anesthetic/surgical technique, and postoperative care will conducted according to institutional protocols; no modifications of any kind will be made for the participants.

SUMMARY:
Introduction: Postoperative atrial fibrillation is one of the most frequent complications in cardiac surgery, with an expected incidence of more than 50% following valve surgery. Hypomagnesemia is also likely to be observed in the postoperative period, and several studies have suggested that it could be related to the incidence of postoperative atrial fibrillation. In this study, via a prospective design and adjustment for multiple covariates, the investigators will seek to determine whether plasma magnesium levels are independently associated with the appearance of postoperative atrial fibrillation.

Methods: An analytical design involving a concurrent cohort will be carried out in a high-complexity hospital with a cardiovascular focus. Serial postoperative plasma magnesium measurements will be included as independent variables in a logistic regression model to determine their association with atrial fibrillation after adjusting for multiple covariates.

ELIGIBILITY:
Inclusion Criteria:

* Adults in postoperative cardiac surgery

Exclusion Criteria:

* Preoperative atrial fibrillation
* Without complete information regarding plasmatic magnesium postoperative measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent cardiac surgery at Fundación Cardioinfantil-Instituto de Cardiología, from May 2015 to May 2016.
Sampling Method: Non-Probability Sample
Enrollment: 435 (Actual)
Dates: Start 2015-05-04 (Actual); Primary Completion 2016-06-03 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Postoperative Atrial fibrilation | Measurement was performed first day after surgery up to 30 days postoperatively or discharge (whichever came first)
  Defined as irregular QRS without p wave during 30 seconds in a 12 derivations EKG.

SECONDARY OUTCOMES:
Mortality | Measurement was performed first day after surgery up to 30 days postoperatively or discharge (whichever came first)
  Overall mortality rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Cardioinfantil-Instituto de Cardiología, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: Undecided
Data from the study would be provided by request to the principal investigator.